CLINICAL TRIAL: NCT01326793
Title: Internet-Based Depression Screening for College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Albert Yeung, Albert Yeung, MD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2008P001438
Record Dates: First submitted 2011-03-25; First posted 2011-03-31 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Major Depressive Disorder
Keywords: telepsychiatry; MDD; Depression; Major Depressive Disorder; Skype; college; university
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Skype Consultation — One-hour Skype consultation with MA-licensed psychiatrist and a written summary of findings.

SUMMARY:
This study aims to determine whether using telecommunication tools, specifically web pages containing online screening instruments and real-time video chat, will be an efficient way to implement Major Depressive Disorder screening among college students. The study also aims to determine if proactive depression screening and free online consultation with a psychiatrist will increase the rate of help-seeking among college students with MDD.

Eligible participants will complete a demographics survey and depression screening assessment online. Those subjects who express suicidality or depressive symptoms will be offered the opportunity to complete a one-time psychiatric consultation with Skype video-conferencing.

ELIGIBILITY:
Inclusion criteria:

* All who consider themselves current undergraduate from Massachusetts colleges are encouraged to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1900 (Actual)
Dates: Start 2008-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
9-item Patient Health Questionnaire | Baseline, Week 8
  Subjects are given the PHQ-9 at baseline, and a 8-week follow-up survey that includes PHQ-9 and questions inquiring whether subject has begun treatment for MDD and whether they faced obstacles in seeking treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Yeung, MD, ScD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Depression Clinical and Research Program at Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Shyu I, Soo JY, Fava M, Kvedar J, Yeung A. Internet Based Depression Screening for College Students. Proceedings of the 163rd Annual Meeting of the American Psychiatric Association (APA). New Orleans, LA, 2010.
- [Result] Soo JY, Shyu, I, Kvedar J, Fava M, Yeung A. The use of Facebook to advertise depression screening among college students: A feasibility and effectiveness study. Proceedings of the 62nd Annual Meeting of the Institute of Psychiatric Services (IPS). Boston, MA, 2010.